CLINICAL TRIAL: NCT00031070
Title: Augmenting the Magnitude of HAART-Induced Immune Restoration With the Use of Cyclosporine
Brief Title: Increasing HAART-Induced Immune Restoration With Cyclosporine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5138; AACTG A5138; ACTG A5139s; AACTG A5139s
Record Dates: First submitted 2002-02-20; First posted 2002-02-22 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2006-08

CONDITIONS: HIV Infections
Keywords: Zidovudine; CD4 Lymphocyte Count; Lamivudine; Cyclosporine; Hepatitis A Vaccine; Rabies Vaccine; abacavir; Antiretroviral Therapy, Highly Active; efavirenz; Treatment Naive
MeSH Terms: conditions — HIV Infections; Hepatitis | interventions — abacavir; Lamivudine; Zidovudine; Cyclosporine; Hepatitis A Vaccines; efavirenz; Heptavalent Pneumococcal Conjugate Vaccine; Rabies Vaccines

INTERVENTIONS:
Drug: Abacavir sulfate, Lamivudine and Zidovudine
Drug: Cyclosporine
Biological: Hepatitis A Vaccine (Inactivated)
Drug: Efavirenz
Biological: Pneumococcal Conjugate Vaccine, Heptavalent
Biological: Rabies Vaccine

SUMMARY:
The purpose of this study is to see if cyclosporine, taken when a patient begins highly active antiretroviral therapy (HAART), increases the number of CD4 T-cells (blood cells that fight infection) in a patient's blood. This study also will explore the safety of briefly giving cyclosporine to patients starting HAART.

DETAILED DESCRIPTION:
The availability of HAART has substantially decreased the morbidity and mortality caused by HIV-1 infection. There is clinical and laboratory evidence suggesting that treatment of HIV-1 infection not only arrests the progressive immune deterioration caused by HIV-1, but also is associated with at least partial immune reconstitution. After starting HAART, most patients with chronic HIV-1 infection experience an increase in CD4 T-cells, but the magnitude of CD4 lymphocyte rise is highly variable. Patients who do not experience a substantial rise in circulating CD4 lymphocytes remain at risk for opportunistic infections. Strategies to enhance immune restoration in HIV-1 disease are needed. Studies have shown that immune restoration after HAART in patients with chronic HIV-1 infection is incomplete. There are, however, several potential methods that can be used that possibly may enhance the magnitude of CD4 lymphocyte rise induced by HAART. It is proposed that the lymphoid tissues, in which lymphocytes are trapped and activated to die, are a major site of immunopathology and cellular losses in HIV-infection. Interference with lymphocyte trapping and death in lymphoid tissues when cyclosporine, an immunosuppressant, is administered at the time of initiation of HAART may result in an enhancement of the magnitude of cellular restoration in patients who initiate HAART.

Patients are randomized to 1 of 2 treatment arms:

Arm A: Weeks 1 to 2: abacavir (ABC)/lamivudine (3TC)/zidovudine (ZDV). Weeks 3 to 48: ABC/3TC/ZDV and efavirenz (EFV).

Arm B: Weeks 1 to 2: ABC/3TC/ZDV and cyclosporine. Weeks 3 to 48: ABC/3TC/ZDV and EFV.

Patients in both arms receive the following immunizations: Weeks 8 and 12: Hepatitis A vaccine inactivated and rabies vaccine.

Week 16: Rabies vaccine. To ascertain whether the augmentation in the rise in CD4 lymphocytes is sustained, the number of circulating CD4 lymphocytes 48 weeks after starting therapy is compared. To examine the functional significance of the cellular increases, the ability of patients to respond to immunization with recall and neoantigens are compared between the cyclosporine plus HAART arm and the HAART alone arm.

Substudy A5139: A 2-week substudy designed to explore the mechanisms of first-phase cellular restoration is performed. Patients undergo 4 lymph node aspirates. Lymphocytes are analyzed by the use of flow cytometry and correlated with findings in the main study. There is no limit on patient enrollment. Patients register to the substudy immediately after randomizing to the main study.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV infected.
* Have received no more than 7 days of any anti-HIV treatment prior to study entry and not within 3 weeks of study entry.
* Have a CD4 cell count greater than 100 cells/mm3 within 30 days prior to study entry.
* Have a viral load greater than 5000 copies/ml within 30 days prior to study entry.
* Agree not to become pregnant or to impregnate during the study. The female/male partners must use 2 acceptable methods of contraception while receiving drugs and for 6 weeks after stopping the study drugs. Women and men who cannot have children do not need to use contraception.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have an AIDS-related infection or abnormal tissue growth within 1 year of study entry.
* Are pregnant or breast-feeding.
* Weigh less than 88 lbs (40 kg).
* Have taken 3TC or nonnucleoside reverse transcriptase inhibitors (NNRTIs).
* Have continuously taken for longer than 3 days any of the following prohibited drugs within 14 days before study entry: angiotensin-converting inhibitors, antibiotics, anticonvulsants, antihistamines, antineoplastics, antifungals, anti-inflammatory drugs, benzodiazepines, calcium channel blockers, gastrointestinal agents, systemic glucocorticoids, immunosuppressives, immunomodulators, potassium-sparing diuretics, statins, allopurinol, amiodarone, bromocryptine, danazol, digoxin, methotrexate, metoclopramide, octreotide, ticlopidine, orlistat, pimozide, nefazodone, fluvoxamine, and ergot derivatives.
* Have taken St. John's wort, grapefruit, or grapefruit juice continuously for longer than 3 days within 14 days before study entry.
* Are allergic or sensitive to study HAART or cyclosporine.
* Abuse drugs or alcohol.
* Have autoimmune disease requiring immunosuppression.
* Have kidney disease or insufficiency.
* Have uncontrolled hypertension.
* Have migraines that require current continuous use of drugs.
* Have a seizure disorder that requires continuous use of anti-seizure drugs.
* Have an HLA B-57 haplotype (this gene has been associated with an increased chance for developing an allergic reaction to ABC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lederman, M.D., Study Chair — Case Western Reserve University
Locations (15):
- United States (15):
  - University of California , Davis Medical Center, Sacramento, California
  - University of Miami, Miami, Florida
  - Rush Presbyterian - Saint Luke's Med Ctr / Infect Dis, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Univ of Minnesota, Minneapolis, Minnesota
  - Washington Univ (St. Louis), St Louis, Missouri
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of North Carolina / Infectious Disease Division, Chapel Hill, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas

REFERENCES:
- [Derived] Lederman MM, Smeaton L, Smith KY, Rodriguez B, Pu M, Wang H, Sevin A, Tebas P, Sieg SF, Medvik K, Margolis DM, Pollard R, Ertl HC, Valdez H. Cyclosporin A provides no sustained immunologic benefit to persons with chronic HIV-1 infection starting suppressive antiretroviral therapy: results of a randomized, controlled trial of the AIDS Clinical Trials Group A5138. J Infect Dis. 2006 Dec 15;194(12):1677-85. doi: 10.1086/509261. Epub 2006 Nov 2. PMID 17109339